CLINICAL TRIAL: NCT02223338
Title: Conjunctival Floral Resistance in a Single Practice Site Comparing Povidone- Iodine Prep With or Without Post-Intravitreal Injection Second Generation Fluoroquinolones.
Brief Title: Bacterial Resistance in Patients Receiving Post-Intravitreal Injection Antibiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, David Sierpina, MD, Loma Linda University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 5140215
Record Dates: First submitted 2014-07-28; First posted 2014-08-22 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Bacterial Resistance
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprofloxacin (Active Comparator): Ciprofloxacin:
  Patients with choroidal neovascularization due to wet age-related macular degeneration or any other cause, clinically significant macular edema or cystoid macular edema over age 18 who have been treated with at least 3 monthly intravitreal injections of an anti-Vascular Endothelial Growth Factor (anti-VEGF) agent in the last 6 months. These patients must have been instructed to use post-injection topical ciprofloxacin 0.3% 4x daily for 3 days. On the visit of their next injection, a conjunctival swab will be taken in the inferior fornix prior to instillation of any ophthalmic drops.
  Interventions: Drug: Ciprofloxacin
- Standard Aseptic Technique (Active Comparator): Standard Aseptic Technique:
  Patients with choroidal neovascularization due to wet age-related macular degeneration or any other cause, clinically significant macular edema or cystoid macular edema over age 18 who have been treated with at least 3 monthly intravitreal injections of an anti-Vascular Endothelial Growth Factor (anti-VEGF) agent in the last 6 months. These injections must have been given with povidone-iodine only applied to the injection site and conjunctival fornix prior to injection, but no post-injection antibiotics were given. On the visit of their next injection, a conjunctival swab will be taken in the inferior fornix prior to instillation of any ophthalmic drops.
  Interventions: Drug: Standard Aseptic Technique

INTERVENTIONS:
Drug: Ciprofloxacin — Use of topical ciprofloxacin 4x daily for 3 days after intravitreal injection using standard aseptic techniques with Povidone-Iodine is a common practice intervention in the United States, and is thought by some to reduce the risk of post-injection endophthalmitis.
  Other Names: ciloxan
  Arms: Ciprofloxacin
Drug: Standard Aseptic Technique — Patients in this group will have received Povidone-Iodine Only following injections of anti-VEGF agents at least 3 times in the last 6 months.
  Other Names: betadyne
  Arms: Standard Aseptic Technique

SUMMARY:
1. Background: Over 1 million intravitreal injections are performed annually in the United States. The most devastating complication related to these injections is endophthalmitis, with an incidence of 0.02 - 0.1% per injection. Techniques aimed at prevention of this complication have been studied, though emergence rates of antibiotic resistant bacteria in a single clinic population comparing antiseptic technique with iodine vs. use of post-injection second generation fluoroquinolones has not been reported in the literature.
2. Objectives: The purpose of the study is to help determine the best way to prevent infection and limit antibiotic resistance in patients receiving eye injections.
3. Procedures Involved (Research Interventions): After the patient is chosen based on inclusion criteria and agrees to participate in the study, exclusion criteria will be reviewed, cognizance will be determined, informed consent and HIPAA compliance forms will be signed. At this point and prior to the instillation of ophthalmic medications, a Rayon swab will be passed along the inferior fornix of the study eye while the patient looks up and the examiner lowers the lower eyelid. The swab will then be used to inoculate chocolate agar and a blood agar culture plates and a glass slide. These will be brought to the FMO microbiology department for culture and Gram stain. All Staphylococcus aureus and coagulase negative Staphylococcus species identified will be subjected to sensitivity testing using the Gram Positive antibiotic panel available at Loma Linda, with the addition of ciprofloxacin.

DETAILED DESCRIPTION:
Previous studies have demonstrated that bacteria in the eye may become resistant to antibiotics used after injections when compared to the bacteria found in untreated eyes. However, no study published to date compares resistance rates in eyes where an iodine-based preparation is used, which is standard of care, to those in which an antibiotic is also given after the injection in a single practice setting. This is an important issue, because resistant bacteria can cause infections that are more damaging and difficult to treat than non-resistant bacteria. Moreover, previous studies have focused on the emergence of resistance to fourth generation fluoroquinolones including moxifloxacin and gatifloxacin, though use of second generation fluoroquinolones is still practiced in the United States by some retina specialists, including at the investigators institution. Currently in the United States, 81% of retina specialists give antibiotics after eye injections, although the results of several large studies suggest that this practice does not reduce rates of endophthalmitis compared with use of iodine alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with choroidal neovascularization due to wet age-related macular degeneration or any other cause, clinically significant macular edema or cystoid macular edema over age 18 who have been treated with at least 3 monthly intravitreal injections of an anti-Vascular Endothelial Growth Factor (anti-VEGF) agent in the last 6 months. These injections must have been given in either Dr. Fan's clinic using povidone-iodine and post-injection topical ciprofloxacin 0.3% 4x daily for 3 days, or in Dr. Rauser's clinic where povidone-iodine only is applied to the injection site and conjunctival fornix but no post-injection antibiotics are given.

Exclusion Criteria:

* Administration of anti-VEGF agents outside of Dr. Fan's or Dr. Rauser's clinics
* Intraocular surgery
* Use of topical antibiotics other than ciprofloxacin 0.3%
* Infections of the eye or ocular adnexa within the last 3 months
* Use of oral antibiotics within the last 30 days
* Contact lens wear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rauser, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University of Health Sciences Faculty Medical Offices, Loma Linda, California, United States

REFERENCES:
- [Background] McCannel CA. Meta-analysis of endophthalmitis after intravitreal injection of anti-vascular endothelial growth factor agents: causative organisms and possible prevention strategies. Retina. 2011 Apr;31(4):654-61. doi: 10.1097/IAE.0b013e31820a67e4. PMID 21330939
- [Background] Moshfeghi AA, Rosenfeld PJ, Flynn HW Jr, Schwartz SG, Davis JL, Murray TG, Smiddy WE, Berrocal AM, Dubovy SR, Lee WH, Albini TA, Lalwani GA, Kovach JL, Puliafito CA. Endophthalmitis after intravitreal vascular [corrected] endothelial growth factor antagonists: a six-year experience at a university referral center. Retina. 2011 Apr;31(4):662-8. doi: 10.1097/IAE.0b013e31821067c4. PMID 21836400
- [Background] Kim SJ, Toma HS. Ophthalmic antibiotics and antimicrobial resistance a randomized, controlled study of patients undergoing intravitreal injections. Ophthalmology. 2011 Jul;118(7):1358-63. doi: 10.1016/j.ophtha.2010.12.014. Epub 2011 Mar 21. PMID 21420176
- [Background] Kim SJ, Toma HS. Antimicrobial resistance and ophthalmic antibiotics: 1-year results of a longitudinal controlled study of patients undergoing intravitreal injections. Arch Ophthalmol. 2011 Sep;129(9):1180-8. doi: 10.1001/archophthalmol.2011.213. PMID 21911665
- [Background] Mino De Kaspar H, Hoepfner AS, Engelbert M, Thiel M, Ta CN, Mette M, Schulze-Schwering M, Grasbon T, Sesma-Vea B, Casas JM, Iturralde-Goni R, Klauss V, Kampik A. Antibiotic resistance pattern and visual outcome in experimentally-induced Staphylococcus epidermidis endophthalmitis in a rabbit model. Ophthalmology. 2001 Mar;108(3):470-8. doi: 10.1016/s0161-6420(00)00545-5. PMID 11237900
- [Background] Miller D, Flynn PM, Scott IU, Alfonso EC, Flynn HW Jr. In vitro fluoroquinolone resistance in staphylococcal endophthalmitis isolates. Arch Ophthalmol. 2006 Apr;124(4):479-83. doi: 10.1001/archopht.124.4.479. PMID 16606872
- [Background] Green-Simms AE, Ekdawi NS, Bakri SJ. Survey of intravitreal injection techniques among retinal specialists in the United States. Am J Ophthalmol. 2011 Feb;151(2):329-32. doi: 10.1016/j.ajo.2010.08.039. Epub 2010 Dec 18. PMID 21168821
- [Background] Bhatt SS, Stepien KE, Joshi K. Prophylactic antibiotic use after intravitreal injection: effect on endophthalmitis rate. Retina. 2011 Nov;31(10):2032-6. doi: 10.1097/IAE.0b013e31820f4b4f. PMID 21659941
- [Background] Cheung CS, Wong AW, Lui A, Kertes PJ, Devenyi RG, Lam WC. Incidence of endophthalmitis and use of antibiotic prophylaxis after intravitreal injections. Ophthalmology. 2012 Aug;119(8):1609-14. doi: 10.1016/j.ophtha.2012.02.014. Epub 2012 Apr 4. PMID 22480743

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciprofloxacin: Ciprofloxacin:
  Patients with choroidal neovascularization due to wet age-related macular degeneration or any other cause, clinically significant macular edema or cystoid macular edema over age 18 who have been treated with at least 3 monthly intravitreal injections of an anti-Vascular Endothelial Growth Factor (anti-VEGF) agent in the last 6 months. These patients must have been instructed to use post-injection topical ciprofloxacin 0.3% 4x daily for 3 days. On the visit of their next injection, a conjunctival swab will be taken in the inferior fornix prior to instillation of any ophthalmic drops.
  Ciprofloxacin: Use of topical ciprofloxacin 4x daily for 3 days after intravitreal injection using standard aseptic techniques with Povidone-Iodine is a common practice intervention in the United States, and is thought by some to reduce the risk of post-injection endophthalmitis.
- Standard Aseptic Technique: Standard Aseptic Technique:
  Patients with choroidal neovascularization due to wet age-related macular degeneration or any other cause, clinically significant macular edema or cystoid macular edema over age 18 who have been treated with at least 3 monthly intravitreal injections of an anti-Vascular Endothelial Growth Factor (anti-VEGF) agent in the last 6 months. These injections must have been given with povidone-iodine only applied to the injection site and conjunctival fornix prior to injection, but no post-injection antibiotics were given. On the visit of their next injection, a conjunctival swab will be taken in the inferior fornix prior to instillation of any ophthalmic drops.
  Standard Aseptic Technique: Patients in this group will have received Povidone-Iodine Only following injections of anti-VEGF agents at least 3 times in the last 6 months.
Period: Overall Study
Arm/Group | Ciprofloxacin | Standard Aseptic Technique
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin | Standard Aseptic Technique | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 12 | 31
  >=65 years | 41 | 48 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.78 (12.99) | 74.68 (13.96) | 72.23 (13.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Resistance of Ocular Flora to Commonly Used Post-injection Prophylactic Antibiotics
Description: Resistance of all coagulase negative staph and staph aureus species to a panel of commonly used antibiotics will be determined and compared between groups. Resistance will be measured using minimum inhibitory concentrations which will be tested on the Siemens MicroScan instrument by doubling broth dilutions. Antibiotic susceptibility interpretations using the categories "S" for susceptible, "I" for Intermediate and "R" for Resistance based on the Clinical and Laboratory Standards Institute (CLSI) guidelines.
  Ciprofloxacin will be tested using the Biomerieux "E test" strip. The test directly quantifies antimicrobial susceptibility in terms of discrete MIC values on a continuous gradient strip. The MIC values are also based on the CLSI guidelines giving interpretations of "S", "I" or "R".
  For information on other antibiotics to be tested, please contact the investigator or provide more characters for input.
Time Frame: Cultured organisms will be subjected to resistance panels once they have grown and been identified. Cultures will be followed for 7 days total, and if no growth is recorded at that time they will be considered sterile.
Population: All culture positive samples growing Staphylococcus aureus or coagulase negative Staphylococcus species.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Standard Aseptic Technique
Number analyzed (Participants) | 18 | 22
Participants | 10 | 6

2. Secondary Outcome: Average Number of Antibiotics to Which Isolated Organisms Were Resistant
Description: Average number of antibiotics to which isolated organisms were resistant, isolated organisms include only coagulase negative Staphylococcus species and Staphylococcus aureus. Antibiotics are those described in the methods section.
Time Frame: Through study completion, average of 4 weeks
Population: All isolates of coagulase negative Staphylococcus and Staphylococcus aureus
Measure: Mean (Standard Deviation); unit: antibiotics
Arm/Group | Ciprofloxacin | Standard Aseptic Technique
Number analyzed (Participants) | 18 | 22
antibiotics | 5.44 (4.29) | 3.23 (3.66)

ADVERSE EVENTS:
Time Frame: 1 week
Description: Data was collected on patients returning to clinic with complaints relating to the study procedure of collecting a conjunctival swab.
Arm/Group | Ciprofloxacin | Standard Aseptic Technique
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes